CLINICAL TRIAL: NCT04216485
Title: Intensive Lifestyle Intervention on Gestational Weight Gain and Development of Gestational Diabetes Mellitus in Overweight/Obese Pregnant Women With a History of Polycystic Ovarian Syndrome
Brief Title: Lifestyle Intervention in Pregnant Women With PCOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Guanghui Li, Associate Professor, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Z161100000516160; Z16110700050000 (Other: Beijing Municipal Science and Technology Commission)
Record Dates: First submitted 2016-11-21; First posted 2020-01-02 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Polycystic Ovary Syndrome; Overweight and Obesity; Gestational Diabetes
MeSH Terms: conditions — Polycystic Ovary Syndrome; Overweight; Obesity; Diabetes, Gestational | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifestyle intervention (Experimental): Intervention group: Intensive lifestyle intervention will be initiated from the first trimester (8-12wks) to delivery, with follow up every 2-4 weeks. Participants in the intervention group will be provided with an individualized dietary protocol with not less than 1500 calories per day in the first trimester and not less than 1800 calories per day after 13 weeks of gestation. Guidance on regular exercise is reinforced at the first and each follow up visit.
  Interventions: Behavioral: Intensive Lifestyle Intervention
- Standard Care (Active Comparator): Standard care group: Participants will receive a 1.5-hour group session in which standard prenatal intervention on diet, nutrition and physical activity and recommendation for gestational weight gain are reviewed by a registered dietitian. Thereafter, participants will receive their regularly scheduled follow up visits without additional lifestyle guidance.
  Interventions: Behavioral: Standard Care

INTERVENTIONS:
Behavioral: Intensive Lifestyle Intervention — Dietary intervention combined with healthy lifestyle counseling
  Arms: Lifestyle intervention
Behavioral: Standard Care — Standard prenatal care on diet, nutrition and physical activity
  Arms: Standard Care

SUMMARY:
Polycystic ovarian syndrome (PCOS) is the most common reproductive disorder in women of childbearing age and is also associated with metabolic abnormalities including obesity, type 2 diabetes, dyslipidemia, etc. Importantly, a number of adverse outcome are seen in pregnancies complicated by PCOS, including gestational diabetes mellitus (GDM), preeclampsia and miscarriage. However, optimal management of PCOS complicated pregnancy is not known. This study seeks to explore whether healthy lifestyle intervention in overweight/obese pregnant women with PCOS could reduce gestational weight gain (GWG) and incidence of GDM.

DETAILED DESCRIPTION:
A randomized controlled trial in PCOS pregnant women will be initiated at 8-12 weeks of gestation util delivery. Participants will be randomly assigned to the control group (standard care) or the intervention group (intensive lifestyle intervention). The intervention will focus on restricting energy intake combined with behavioral lifestyle modification through participation in group sessions and individual counseling. The primary outcome will be GWG and secondary outcome will be the incidence of GDM.

Our hypothesis is that intensive lifestyle intervention in overweight/obese pregnant women with PCOS will decrease GWG and reduce the incidence of GDM.

ELIGIBILITY:
Inclusion Criteria:

* gestational age between 8 and 12 weeks of gestation, pre-pregnancy BMI≥25 (kg/m2)
* age ≥18 years, and a singleton pregnancy.

Exclusion Criteria:

* patients with prediabetes and diabetes, hypertension, chronic renal disease, thyroid disorder
* gestational weeks ≥ 13
* age <18 years
* multiple pregnancy
* uterine malformation
* or physical restriction that prevents exercise.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 296 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Gestational weight gain | From date of randomization until the date of delivery, assessed up to 9 months

SECONDARY OUTCOMES:
Incidence of Gestational Diabetes Mellitus | From enrollment to 24-28 weeks of gestation

CONTACTS AND LOCATIONS:
Overall Officials: Guanghui Li, MD, PhD, Principal Investigator — Beijing Obstetrics and Gynecology Hospital
Locations (1):
- Beijing Obstetrics and Gynecology Hospital,Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No